CLINICAL TRIAL: NCT06343649
Title: Response in Patients with Persistent Pelvic Pain to Explicit Motor Imagery Through Auditory or Visual Input
Brief Title: Response in Patients with Persistent Pelvic Pain to Motor Imagery Through Auditory or Visual Input. a Pilot Randomized Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Lecturer PhD. Departament of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEUMA 187-2023-H
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Pain
Keywords: pain; pelvic pain
MeSH Terms: conditions — Pelvic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual Explicit Motor Imagery (Experimental): 6 exercises of Explicit Motor Imagery, administered on alternate days, using visual inputs in the form of images.
  Interventions: Other: Visual
- Auditory Explicit Motor Imagery (Experimental): 6 exercises of Explicit Motor Imagery, administered on alternate days, using auditory inputs in the form of audio recordings.
  Interventions: Other: Auditory

INTERVENTIONS:
Other: Visual — Delivery of images to conduct several exercises of Explicit Motor Imagery
  Arms: Visual Explicit Motor Imagery
Other: Auditory — Delivery of audio recordings to conduct several exercises of Explicit Motor Imagery
  Arms: Auditory Explicit Motor Imagery

SUMMARY:
The goal of this clinical trial is to compare the response of Explicit Motor Imagery interventions in patients suffering Persistent Pelvic Pain. The main question it aims to answer is:

• Does the modality of application of Explicit Motor Imagery, either through visual or auditory stimuli, influence the response in patients suffering Persistent Pelvic Pain?

Participants will receive an online Explicit Motor Imagery program either through visual inputs or auditory inputs. They will be instructed to follow the program en register their response.

Researchers will compare visual Explicit Motor Imagery and auditory Explicit Motor Imagery to see if different inputs generate different responses in patients suffering Persistent Pelvic Pain.

ELIGIBILITY:
Inclusion Criteria:

* Experience persistent pain for a minimum duration of six months.
* Achieve a minimum score of six points on the Chronic Pelvic Pain Questionnaire (CPPQ), a validated instrument designed to assess the discrimination of pain.

Exclusion Criteria:

* Participants with a medically diagnosed condition that logically accounts for the presence of pain during the aforementioned six-month period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | Baseline to two weeks
  Self-administered scale that requires the patient to rate their pain intensity on a 0-10 scale, where 0 is no pain and 10 is the worst pain imaginable. Higher scores indicate worse outcomes.
Pain Vigilance and Awareness Questionnaire | Baseline to two weeks
  Self-administered questionnaire to measure attention to pain. 16- item questionnaire, where each item is scored as a six- point Likert scale that ranges from zero (never) to five (always), resulting in a sum score between zero and 80. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire-Revised | Baseline
  Assesses visual and kinesthetic movement imagery abilities. Self-adminstered instrument comprised of 2 subscales: Visual Imagery (4 items) and Kinesthetic Imagery (4 items). Respondents assign a value from a 7-point scale, which indicates the ease or difficulty with which the movement was seen/felt. Higher scores indicate worse movement imagery abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Perez-Dominguez B, Arce-Elorza A, Rubio-Garcia I, Diaz-Mohedo E. Response in Patients With Persistent Pelvic Pain to Motor Imagery Through Auditory or Visual Input-A Pilot Randomized Trial. Pain Res Manag. 2025 Feb 10;2025:1412626. doi: 10.1155/prm/1412626. eCollection 2025. PMID 39963311